CLINICAL TRIAL: NCT03768700
Title: Characteristics and Evolution of Hospitalized Patients in Post-Resuscitation Rehabilitation Care Units (SRPR)
Acronym: Cohorte-SRPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17008J; 2018-A00743-52 (Other: ANSM)
Record Dates: First submitted 2018-10-22; First posted 2018-12-07 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Hospitalization in a Post-Resuscitation Rehabilitation Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Hospitalization in a Post-Resuscitation Rehabilitation Care Units (SRPR)
  Interventions: Other: Data gathering

INTERVENTIONS:
Other: Data gathering — Questionnaires and collection of medical data on patients during hospitalization, at D28, at 90 and at 1 year

SUMMARY:
Non-interventional cohort study (on data), prospective national multicenter. Inclusion of patients as they enter in a post-intensive care rehabilitation unit (SRPR) .

Collection of data after inclusion, from patients' records during their stay (weekly follow-up) to the SRPR and at their discharge, to D28, D90 and at 1 year after their hospitalization from hospital reports or call of the attending physician.

DETAILED DESCRIPTION:
For one year, all patients, adults and children hospitalized in a post-intensive care rehabilitation unit (SRPR) of Ile de France and Rouen will be offered to participate in the SRPR Cohort in order to have a completeness of data on a new practice.

The study of these data will make it possible to know the future of the patients and to establish criteria prior to the admission in the SRPR which could make it possible to predict this future and to select the patients as well as possible. It will also make it possible to know the impact of care on the outcome of patients at discharge, at 28 days, 90 days and 1 year of their admission to SRPR to improve practices.

This research will focus on the collection of data from patients' medical records. General information about their stay in the intensive care unit - including the patient's ventilatory status - will be collected upon arrival at the SRPR units, during their stay (weekly follow-up), at the exit of the SRPR, at D28, and in the longer term. (J90 and J365 of the entry into the SRPR unit) where will be listed more comprehensive data with, in addition to general information, data on nutritional, neurological, neuromuscular, respiratory and biological hemodynamic assessments will be collected.

In addition to the common data base, each type of SRPR (respiratory and pediatric neurology) will collect data that is specific to its specialty.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in a Post-Resuscitation Rehabilitation Care Units (SRPR) of Ile de France and Rouen

Exclusion Criteria:

* Refusal of access to the data by the patient or the designated trusted person or the holder (s) of parental authority (pediatric population)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalization in a Post-Resuscitation Rehabilitation Care Units (SRPR) of Ile de France and Rouen
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation status of patients discharged from SRPR | 28 days
  Describe the ventilatory status of patients hospitalized in SRPR at the SRPR exit: during the week before the evaluation, does the patient use at least one time: invasive or noninvasive ventilation?

SECONDARY OUTCOMES:
Functional status assessed by the functional independence measurement scale (MIF) at entry to the SRPR and weekly follow-up during the stay and discharge of the SRPR, at discharge from the hospital, at Day 28, Day 90 and at 1 year. | one year
  Describe the clinico-biological characteristics of patients prior to admission to SRPRs and their future in order to better select them.
Vital status at the exit of the SRPR at Day 28, Day 90 and at 1 year. The starting point is the entry into the SRPR unit. | Between the exit of the SRPR and up to one year after entry into the SRPR unit
  The only one parameters that we will measure will be vital status: alive or not?
Ventilatory status at discharge from the hospital, Day 28, Day 90 and at 1 year. The starting point is the entry into the SRPR unit. | Between the exit of the SRPR and up to one year after entry into the SRPR unit
  During the week before the evaluation, does the patient use at least one time: invasive or noninvasive ventilation?
Length of stay in intensive care unit, SRPR and hospital | one year
Evaluation of swallowing of patients | one day
  Evaluate by clinical data recorded in the medical file at upon entry into SRPR service.
Evaluation of nutrition of patients | one day
  Evaluate by clinical data recorded in the medical file at upon entry into SRPR service.
Evaluation of nutritional status of patients | one day
  Evaluate by clinical data recorded in the medical file: weight in kilograms, height in meters and a combined BMI= weight/height in kg/m^2) and measurement of albumin (g/l) and measurement of prealbuminemia (g/l) at upon entry into SRPR service.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DEMOULE, Pr, Principal Investigator — Hôpital Pitié-Salpêtrière - AP-HP
Locations (10):
- France (10):
  - Groupe hospitalier des portes de l'Oise, Beaumont-sur-Oise
  - Centre hospitalier de Bligny, Briis-sous-Forges
  - Hôpital d'instruction des armées - Percy, Clamart
  - Hôpital de Forcilles, Férolles-Attilly
  - Hôpital Raymond Poincaré - SRPR pédiatrique, Garches
  - Hôpital Raymond Poincaré de Garches - SRPR neurologique, Garches
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Sainte-Anne, Paris
  - Hôpital Charles-Nicolle - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No